CLINICAL TRIAL: NCT01584752
Title: Clinical Multicenter Study of the Efficacy of Gore-BioA Fistula Plug in High Transsphincteric Perianal Fistulas
Brief Title: Gore-BioA Fistula Plug to Treat Transsphincteric Fistulas
Status: Terminated | Type: Observational
Why Stopped: Recruitment not satisfactory
Sponsor: Central Finland Hospital District (Other)
Responsible Party: Sponsor
Other Study IDs: KSSHP1U/2011
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Anal Fistula; Fecal Incontinence; Surgery
MeSH Terms: conditions — Rectal Fistula; Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fistula patients: Gore-BioA Fistula Plug
  Interventions: Procedure: Gore-BioA Fistula Plug

INTERVENTIONS:
Procedure: Gore-BioA Fistula Plug — Gore-BioA Fistula Plug

SUMMARY:
This is a prospective clinical study on the efficacy of Gore-BioA fistula plug in high transsphincteric fistulas. Follow-up time is six months

DETAILED DESCRIPTION:
Inclusion criteria for the study is a patient with ultrasound or MRI proven high transsphincteric perianal fistula. Patients with Crohns disease, immunosuppressive medication, anovaginal fistula, radiation therapy or chemotherapy are excluded. A Seton is placed in the fistula track for two months before the application of the plug. Patients are followed up for six months. Symptoms of fecal incontinence before and after intervention are monitored with the Cleveland clinic incontinence score.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years, male or female
* High cryptoglandular perianal fistula
* Written approval for the study
* Sufficient co-operation for the study
* Localization of the fistula by ultrasound or MRI

Exclusion Criteria:

* Crohns disease
* Immunosuppressive treatment
* Anovaginal fistula
* Radiation therapy 6 months before study
* Chemotherapy 6 months before study
* Low- or intersphincteric fistula

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inhabitants of Finland
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Healing of the fistula | 6 months

SECONDARY OUTCOMES:
Symptoms of fecal incontinence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matti V Kairaluoma, ph.D, Study Director — Central Hospital, Jyväskylä, Finland
Locations (7):
- Finland (7):
  - Helsinki University Hospital, Helsinki
  - Central Hospital, Joensuu
  - Central Hospital, Jyväskylä
  - Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Central Hospital, Seinäjoki
  - Turku University Hospital, Turku